CLINICAL TRIAL: NCT04818866
Title: The International Study of Inflammation in COVID-19: A Prospective Multi-Center Observational Study Examining the Role of Biomarkers of Inflammation in Predicting Covid-19 Related Outcomes in Hospitalized Patients
Brief Title: International Study of Inflammation in COVID-19
Acronym: ISIC
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Rush University (Other); Copenhagen University Hospital, Hvidovre (Other); University of Athens (Other); Heinrich-Heine University, Duesseldorf (Other); University of Thessaly (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Salim S. Hayek, Assistant Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00178971-a
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Outcome, Fatal; Respiratory Failure; Acute Kidney Injury; Inflammation
Keywords: SuPAR; CRP; D-dimer; Ferritin; Interleukin-6; Procalcitonin; lactate dehydrogenase; biomarkers
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Acute Kidney Injury; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma or serum samples collected within 48 hours of presentation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized for Covid-19
  Interventions: Diagnostic Test: SuPAR, C-reactive protein, Ferritin, D-Dimer, Procalcitonin, Interleukin-6, Lactate Dehydrogenase

INTERVENTIONS:
Diagnostic Test: SuPAR, C-reactive protein, Ferritin, D-Dimer, Procalcitonin, Interleukin-6, Lactate Dehydrogenase — Biomarkers of inflammation

SUMMARY:
This is a prospective multi-center observational study which purpose is to evaluate the ability of blood-based inflammatory markers to risk-stratify patients hospitalized for Covid-19. Blood-based biomarkers examined include: soluble urokinase plasminogen activator receptor (suPAR), C-reactive protein (CRP), procalcitonin, D-dimer, ferritin, lactate dehydrogenase and interleukin-6.

DETAILED DESCRIPTION:
All consecutive patients hospitalized specifically for Covid-19 at the University of Michigan in Ann Arbor from February 1st, 2020 to date are included. Other participating centers will enroll patients depending on their variable capacity. Patients with a positive test for SARS-CoV-2 but hospitalized for non-Covid-19 reasons were excluded. Blood-based biomarkers including soluble urokinase plasminogen activator receptor (suPAR), C-reactive protein (CRP), procalcitonin, D-dimer, ferritin, lactate dehydrogenase and interleukin-6 are measured in samples collected within 48 hours of presentation. The primary outcome of the study is the composite endpoint of in-hospital mortality, need for mechanical ventilation and need for renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 test result
* Covid-19 as the primary reason for hospitalization

Exclusion Criteria:

* Hospitalized primarily for non-Covid-19 reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized primarily for Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 4463 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
In-hospital incidence of death, need for mechanical ventilation and need for renal replacement therapy | during COVID91 related hospitalization, up to 6 months
  Composite outcome of death, need for mechanical ventilation, need for renal replacement therapy

SECONDARY OUTCOMES:
Length of Hospitalization | up to 6 months
  Duration of hospitalization
Acute Kidney Injury | within 6 months
  Per KDIGO criteria
Cardiovascular Events | within 6 months
  In-hospital new diagnosis heart failure, arrhythmia, myocardial infarction
Death | within 6 months
  In-hospital mortality
Need for renal replacement therapy | within 6 months
  In-hospital renal replacement therapy or dialysis
Need for mechanical ventilation | within 6 months
  Respiratory failure requiring mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Salim S Hayek, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Due to consent waiver, individual participant data cannot be shared with investigators outside the University of Michigan

REFERENCES:
- [Background] Rovina N, Akinosoglou K, Eugen-Olsen J, Hayek S, Reiser J, Giamarellos-Bourboulis EJ. Soluble urokinase plasminogen activator receptor (suPAR) as an early predictor of severe respiratory failure in patients with COVID-19 pneumonia. Crit Care. 2020 Apr 30;24(1):187. doi: 10.1186/s13054-020-02897-4. No abstract available. PMID 32354367
- [Background] Azam TU, Berlin H, Anderson E, Pan M, Shadid HR, Padalia K, O'Hayer P, Meloche C, Feroze R, Michaud E, Launius C, Blakely P, Bitar A, Willer C, Pop-Busui R, Carethers JM, Hayek SS. Differences in Inflammation, Treatment, and Outcomes Between Black and Non-Black Patients Hospitalized for COVID-19: A Prospective Cohort Study. Am J Med. 2022 Mar;135(3):360-368. doi: 10.1016/j.amjmed.2021.10.026. Epub 2021 Nov 16. PMID 34793753
- [Background] Vasbinder A, Anderson E, Shadid H, Berlin H, Pan M, Azam TU, Khaleel I, Padalia K, Meloche C, O'Hayer P, Michaud E, Catalan T, Feroze R, Blakely P, Launius C, Huang Y, Zhao L, Ang L, Mikhael M, Mizokami-Stout K, Pennathur S, Kretzler M, Loosen SH, Chalkias A, Tacke F, Giamarellos-Bourboulis EJ, Reiser J, Eugen-Olsen J, Feldman EL, Pop-Busui R, Hayek SS; ISIC Study Group. Inflammation, Hyperglycemia, and Adverse Outcomes in Individuals With Diabetes Mellitus Hospitalized for COVID-19. Diabetes Care. 2022 Mar 1;45(3):692-700. doi: 10.2337/dc21-2102. PMID 35045184
- [Background] Pan M, Vasbinder A, Anderson E, Catalan T, Shadid HR, Berlin H, Padalia K, O'Hayer P, Meloche C, Azam TU, Khaleel I, Michaud E, Blakely P, Bitar A, Huang Y, Zhao L, Pop-Busui R, Loosen SH, Chalkias A, Tacke F, Giamarellos-Bourboulis EJ, Reiser J, Eugen-Olsen J, Hayek SS; ISIC Group. Angiotensin-Converting Enzyme Inhibitors, Angiotensin II Receptor Blockers, and Outcomes in Patients Hospitalized for COVID-19. J Am Heart Assoc. 2021 Dec 21;10(24):e023535. doi: 10.1161/JAHA.121.023535. Epub 2021 Dec 10. PMID 34889102
- [Background] Azam TU, Shadid HR, Blakely P, O'Hayer P, Berlin H, Pan M, Zhao P, Zhao L, Pennathur S, Pop-Busui R, Altintas I, Tingleff J, Stauning MA, Andersen O, Adami ME, Solomonidi N, Tsilika M, Tober-Lau P, Arnaoutoglou E, Keitel V, Tacke F, Chalkias A, Loosen SH, Giamarellos-Bourboulis EJ, Eugen-Olsen J, Reiser J, Hayek SS; International Study of Inflammation in COVID-19. Soluble Urokinase Receptor (SuPAR) in COVID-19-Related AKI. J Am Soc Nephrol. 2020 Nov;31(11):2725-2735. doi: 10.1681/ASN.2020060829. Epub 2020 Sep 22. PMID 32963090
- [Background] Hayek SS, Roderburg C, Blakely P, Launius C, Eugen-Olsen J, Tacke F, Ktena S, Keitel V, Luedde M, Giamarellos-Bourboulis EJ, Luedde T, Loosen SH. Circulating Osteopontin Levels and Outcomes in Patients Hospitalized for COVID-19. J Clin Med. 2021 Aug 30;10(17):3907. doi: 10.3390/jcm10173907. PMID 34501358
- [Background] Vasbinder A, Meloche C, Azam TU, Anderson E, Catalan T, Shadid H, Berlin H, Pan M, O'Hayer P, Padalia K, Blakely P, Khaleel I, Michaud E, Huang Y, Zhao L, Pop-Busui R, Gupta S, Eagle K, Leaf DE, Hayek SS; STOP-COVID Investigatorsdouble dagger. Relationship Between Preexisting Cardiovascular Disease and Death and Cardiovascular Outcomes in Critically Ill Patients With COVID-19. Circ Cardiovasc Qual Outcomes. 2022 Oct;15(10):e008942. doi: 10.1161/CIRCOUTCOMES.122.008942. Epub 2022 Oct 4. PMID 36193749
- [Background] Luo S, Vasbinder A, Du-Fay-de-Lavallaz JM, Gomez JMD, Suboc T, Anderson E, Tekumulla A, Shadid H, Berlin H, Pan M, Azam TU, Khaleel I, Padalia K, Meloche C, O'Hayer P, Catalan T, Blakely P, Launius C, Amadi KM, Pop-Busui R, Loosen SH, Chalkias A, Tacke F, Giamarellos-Bourboulis EJ, Altintas I, Eugen-Olsen J, Williams KA, Volgman AS, Reiser J, Hayek SS; ISIC (International Study of Inflammation in COVID-19) Group. Soluble Urokinase Plasminogen Activator Receptor and Venous Thromboembolism in COVID-19. J Am Heart Assoc. 2022 Sep 20;11(18):e025198. doi: 10.1161/JAHA.122.025198. Epub 2022 Aug 4. PMID 35924778
- [Background] Zhu K, Mukherjee K, Wei C, Hayek SS, Collins A, Gu C, Corapi K, Altintas MM, Wang Y, Waikar SS, Bianco AC, Koch A, Tacke F, Reiser J, Sever S. The D2D3 form of uPAR acts as an immunotoxin and may cause diabetes and kidney disease. Sci Transl Med. 2023 Sep 20;15(714):eabq6492. doi: 10.1126/scitranslmed.abq6492. Epub 2023 Sep 20. PMID 37729431
- [Derived] Chalkias A, Huang Y, Ismail A, Pantazopoulos I, Papagiannakis N, Bitterman B, Anderson E, Catalan T, Erne GK, Tilley CR, Alaka A, Amadi KM, Presswalla F, Blakely P, Bernal-Morell E, Cebreiros Lopez I, Eugen-Olsen J, Garcia de Guadiana Romualdo L, Giamarellos-Bourboulis EJ, Loosen SH, Reiser J, Tacke F, Skoulakis A, Laou E, Banerjee M, Pop-Busui R, Hayek SS; International Study of Inflammation in COVID-19 (ISIC) Investigator Group. Intubation Decision Based on Illness Severity and Mortality in COVID-19: An International Study. Crit Care Med. 2024 Jun 1;52(6):930-941. doi: 10.1097/CCM.0000000000006229. Epub 2024 Feb 23. PMID 38391282